CLINICAL TRIAL: NCT02653456
Title: A Prospective, Multi Center Pilot Study Evaluating Plaque Photoablation Using the RA-308 Excimer Laser in Subjects With Symptomatic Infrainguinal Lower Extremity Vascular Disease
Brief Title: Evaluating Plaque Photoablation Using an Excimer Laser in Patients With Lower Extremity Vascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ra Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMS-102
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Arterial Disease
Keywords: excimer laser; percutaneous catheter; photoablation; chronic total occlusion; symptomatic infrainguinal lower extremity vascular disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (1):
- RA-308 Excimer Laser and DABRA Catheter (Experimental): Treatment with the RA-308 excimer laser and DABRA catheter to treat chronic total occlusions that cannot be crossed with standard guidewires. The catheter and laser are a system, and cannot be used separately.
  Interventions: Device: RA-308 Excimer Laser and DABRA Catheter

INTERVENTIONS:
Device: RA-308 Excimer Laser and DABRA Catheter — See information already included in arm description

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of an excimer laser in the treatment of patients with lower extremity vascular disease with chronic total occlusions.

DETAILED DESCRIPTION:
The study is a multi center, prospective, non-randomized, open-label study conducted at a minimum of one investigational center. 50 subjects can be enrolled. Follow-up occurs at the end of the procedure in the form of an angiogram to determine if the lesion was crossed. Additional follow-up may not necessary because of the binary nature of the crossing, and also because any future follow-up would be assessing the effectiveness of adjunct therapy, e.g. balloon angioplasty. Long term results are entirely dependent on this subsequent treatment. Because the DABRA crosser only allows adjunct devices to be used, 30-day follow-up measuring the performance of the adjunct therapy might affect the physician's choice of therapy, and compromise the patient's treatment. Therefore, 30-day follow-up, which evaluates the effectiveness of the adjunct therapy, might raise ethical concerns. However, the follow-up can be done by Ankle-Brachial Index, Doppler ultrasound, auscultation, or by discussion of the level of claudication and motion pain with the patient. To evaluate the safety and efficacy of the RA-308 Excimer Laser System and DABRA Catheter for treating subjects with symptomatic infrainguinal lower extremity vascular disease with chronic total occlusions that cannot be crossed with standard guide wires, or lesions where an attempt to cross would, in the opinion of the interventionalist, result in either a subintimal path or a perforation.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* symptomatic infrainguinal lower extremity vascular disease (Rutherford category 3, 4, 5 or 6), stable for at least 2 weeks prior to study inclusion
* lesions in the superficial femoral artery (SFA), popliteal, or infrapopliteal arteries at least one angiographically identifiable infrageniculate artery
* patients must be poor surgical candidates, indicated by at least one of the following conditions:
* absence of venous autologous grafts (that is, lack of a suitable vein to use for bypass)
* poor (diffusely diseased or <=1mm diameter) or no distal vessels available for graft anastamosis
* high risk of surgical mortality, evidenced by American Society of Anesthesiologists Physical Class 4 or higher

Exclusion Criteria:

* age below 18 years
* pregnancy, or plan to become pregnant
* participation in another cardiovascular or peripheral vascular study
* myocardial infarction (MI) in prior month
* stents at treatment site
* disorders or allergies precluding use of radiographic contrast
* renal insufficiency sever enough to contraindicate use of radiographic contrast
* contraindication to treatment with anticoagulants
* untreated ipsilateral iliac stenosis >70%
* inability or unwillingness of the patient to comply with intended examinations
* unavailability of required procedural or imaging equipment
* lesion located in a graft
* hemodynamically significant arrhythmia or left ventricular ejection fraction <20%
* life expectancy less than 6 months
* necrosis necessitating major amputation
* unwillingness of the patient to be anti-coagulated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehtisham Mahmud, Principal Investigator — UCSD
Locations (3):
- United States (3):
  - California Heart & Vascular Clinic, El Centro, California
  - University of California San Diego, San Diego, California
  - Merit Health Wesley, Hattiesburg, Mississippi

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- RA-308 Excimer Laser and DABRA Catheter: Treatment with the RA-308 excimer laser and DABRA catheter to treat chronic total occlusions in patients with symptomatic infrainguinal lower extremity vascular disease.
Period: Overall Study
Arm/Group | RA-308 Excimer Laser and DABRA Catheter
Started | 64
Completed | 59
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: subjects have a chronic total occlusion in the infrainguinal lower extremities
Groups:
- RA-308 Excimer Laser and DABRA Catheter: Treatment with the RA-308 excimer laser and DABRA catheter to treat chronic total occlusions in patients with symptomatic infrainguinal lower extremity vascular disease. The catheter and laser are a system, and cannot be used separately.
  RA-308 Excimer Laser and DABRA Catheter: See information already included in arm description
Arm/Group | RA-308 Excimer Laser and DABRA Catheter
Number analyzed (Participants) | 64
Age, Continuous [Mean (Full Range); unit: years] | 72 [47 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 64
Region of Enrollment [Number; unit: participants]
  United States | 49
  Mexico | 15
Chronic total occlusion [Count of Participants; unit: Participants] | 64

OUTCOME MEASURES:

1. Primary Outcome: Crossing the Target Lesion
Description: Crossing the target lesion based on angiographic analysis
Time Frame: at time of procedure
Measure: Count of Participants; unit: Participants
Arm/Group | RA-308 Excimer Laser and DABRA Catheter
Number analyzed (Participants) | 64
Participants | 60

2. Secondary Outcome: Number of Participants With no Device-related Major Adverse Events
Description: Number of participants with no device-related major adverse events as determined by physician evaluation
Time Frame: at time of procedure, up to an hour
Measure: Count of Participants; unit: Participants
Arm/Group | RA-308 Excimer Laser and DABRA Catheter
Number analyzed (Participants) | 64
Participants | 0

3. Secondary Outcome: Number of Participants With Target Lesion Revascularization
Description: Number of participants with target lesion revascularization as determined by physician evaluation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | RA-308 Excimer Laser and DABRA Catheter
Number analyzed (Participants) | 59
Participants | 0

4. Secondary Outcome: Number of Participants With Target Lesion Revascularization
Description: Number of participants with target lesion revascularization as determined by physician evaluation
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RA-308 Excimer Laser and DABRA Catheter
Number analyzed (Participants) | 38
Participants | 0

ADVERSE EVENTS:
Time Frame: adverse event data was collected from the time of the procedure up to 6 months post-procedure
Arm/Group | RA-308 Excimer Laser and DABRA Catheter
All-Cause Mortality (participants affected / at risk) | 0/64
Serious Adverse Events (participants affected / at risk) | 0/64
Other Adverse Events (participants affected / at risk) | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT02653456/Prot_SAP_002.pdf